CLINICAL TRIAL: NCT07007299
Title: Safety and Efficacy of Integrative Korean Medicine Treatment for Elderly After Traffic Accident: Retrospective Chart Review Study
Brief Title: Safety and Efficacy of Integrative Korean Medicine Treatment for Elderly After Traffic Accident
Status: Recruiting | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: JS-CT-2024-07
Record Dates: First submitted 2025-04-25; First posted 2025-06-05 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Musculoskeletal Diseases or Conditions; Traffic Accident; Elderly (People Aged 65 or More)
Keywords: pharmacopuncture; herbal medicine; elderly; korean medicine; complementary and alternative medicine; acupuncture
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study was to analyze the medical records of elderly traffic accident patients hospitalized at 4 branches of Jaseng Korean Medicine Hospital to determine the status of elderly patients and the effectiveness and safety of Korean medicine combination treatment.

DETAILED DESCRIPTION:
This study was retrospective chart review study and was conducted in 4 branches of Jaseng Korean Medicine Hospital (Gangnam, Bucheon, Daejeon, Haeundae).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years or older at the time of first visit
* Patients who visited our hospital due to symptoms caused by a traffic accident and received integrated oriental medicine treatment at least once as an inpatient treatment

Exclusion Criteria:

* If only consultation was conducted at the hospital or only Western medicine treatment was conducted
* If only outpatient treatment was received without hospitalization
* If other researcher judges that participation in the study is difficult

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: From January 1, 2021 to December 31, 2023, only patients aged 65 years or older who visited the four branches of Jaseng Oriental Hospital (Gangnam, Bucheon, Daejeon, Haeundae) and received inpatient treatment after being injured in a traffic accident and who meet the selection criteria are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | The results are measured for each patient at admission (before) and discharge (after) from January 2021 to December 31, 2023.
  NRS uses an 11-point scale to evaluate current main pain and radiating pain where no pain is indicated by '0', and the worst pain imaginable by '10'.

SECONDARY OUTCOMES:
euroqol-5 dimension (EQ-5D) | The results are measured for each patient at admission (before) and discharge (after) from January 2021 to December 31, 2023.
  EQ-5D is most widely used as a method of indirectly calculating the quality of life from various aspects. The EQ-5D consists of 5 questions (mobility, self-care, usual activities, pain, anxiety/depression) that ask about the current state of health, and answers each question with 5 likert. (1=I have no problems about, 2=I have slight problems about, 3=I have moderate problems about, 4=I have severe problems about, 5=I am unable to about).
Neck Disability Index (NDI) | The results are measured for each patient at admission (before) and discharge (after) from January 2021 to December 31, 2023.
  NDI is a functional disability questionnaire. The possible range of each item score is 0 to 5. Total score range is 0 (better outcome) to 100 (worse outcome).
Oswestry Disability Index (ODI) | The results are measured for each patient at admission (before) and discharge (after) from January 2021 to December 31, 2023.
  ODI is a 10-item questionnaire developed to evaluate the degree of disability for lower back pain. Each item is divided into 6 levels, and 0 to 5 points are awarded. The higher the score, the greater the degree of disability.
Adverse Events (AE) | The period of hospitalization is limited to January 2021 to December 2023.
  All adverse events complained of by the patient during the period of hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, Ph.D, Study Director — Jaseng Medical Foundation
Locations (4):
- South Korea (4):
  - Daejeon Jaseng Hospital of Korean Medicine, Daejeon, Daejeon
  - Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu
  - Bucheon Jaseng Hospital of Korean Medicine, Bucheon-si, Gyeonggi-do
  - Haeundae Jaseng Hospital of Korean Medicine, Busan

REFERENCES:
- [Derived] Shin JY, Lee YS, Lee SH, Noh JH, Lee YJ, Ha IH, Lee SW. Real-world evidence on the safety and effectiveness of integrative Korean medicine for older patients post-traffic accident: A retrospective observational study. Medicine (Baltimore). 2025 Nov 28;104(48):e46144. doi: 10.1097/MD.0000000000046144. PMID 41327701